CLINICAL TRIAL: NCT02983851
Title: Initial Ventilation Strategy for Adult Immunocompromised Patients With Acute Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Ministry of Health, China (Other Government); Fujian Provincial Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Renmin Hospital of Wuhan University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); General Hospital of Ningxia Medical University (Other); Tianjin Medical University General Hospital (Other); Second Xiangya Hospital of Central South University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Cangzhou Central Hospital (Other); Handan First Hospital (Other)
Responsible Party: Principal Investigator, Yi Li, MD, Chief physician of Emergency Department, professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VENIM
Record Dates: First submitted 2016-11-25; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Immunocompromised Patients; Acute Respiratory Failure
Keywords: Noninvasive mechanical ventilation; Invasive mechanical ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noninvasive mechanical ventilation (Experimental): Patients in this group will receive Noninvasive mechanical ventilation as the initial mechanical ventilation (MV) strategy, irrespective of whether Invasive mechanical ventilation is used later during the following treatment.
  Interventions: Procedure: Noninvasive mechanical ventilation
- Invasive mechanical ventilation (Active Comparator): Patients in this group will receive Invasive mechanical ventilation as the initial MV strategy, irrespective of whether Noninvasive mechanical ventilation is used later during the following treatment.
  Interventions: Procedure: Invasive mechanical ventilation

INTERVENTIONS:
Procedure: Noninvasive mechanical ventilation — Noninvasive mechanical ventilation will be delivered to the patient through a mask. The mask will be adjusted and connected to a ventilation system.
  Arms: Noninvasive mechanical ventilation
Procedure: Invasive mechanical ventilation — Invasive mechanical ventilation will be initially performed by using the volume controlled mode, and could be adjusted to pressure controlled mode or other modes based on clinical situation.
  Arms: Invasive mechanical ventilation

SUMMARY:
VENIM is a multicenter, open-label, parallel-group randomized controlled trial of studying the initial ventilation strategy for adult immunocompromised patients with acute respiratory failure.

DETAILED DESCRIPTION:
The VENIM is a multicenter randomized controlled trial (RCT) comparing the effects of NIV compared with IMV in adult immunocompromised patients with moderate to severe acute respiratory failure (ARF). Patients who meet the indications for both ventilatory supports will be included. The intervention will consist of randomly allocation, treatment with NIV or IMV, concomitant medication. Primary outcome is 30-day hospital mortality. Secondary outcomes include in-hospital mortality, length of stay in hospital, improvement of oxygenation, nosocomial infections, seven-day organ failure, adverse events of intervention, et al. Subgroups with different disease severity, causes of immunodeficiency and types of ARF will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years old ≤ age ≤ 80 years old) immunocompromised patients admitted to hospital with moderate to severe ARF diagnosed within the last 72 hours, which meets the indications for ventilatory support.
* Patients are considered as moderate to severe ARF when the ratio of the partial pressure of arterial oxygen to the fraction of inspired oxygen (PaO2/FiO2) is between 85 and 170 while the patient is breathing oxygen through a Venturi mask, or clinically diagnosed as the following:

  1. 30 mmHg < PaO2 < 50 mmHg on room air;
  2. Clinical evidence of respiratory distress (intercostal recession, polypnea >35/min or dyspnea at rest).
* Patients are considered as immunocompromised when clinically diagnosed as at least one of the following:

  1. HIV infection;
  2. Hematologic malignancy or solid tumor under chemotherapy;
  3. Solid organ or stem cell transplant;
  4. Long-term (>30 days) or high dose steroids (>1 mg/kg/d prednisone equivalent) usage and/or any other immunosuppressive drugs;
  5. Neutropenia (defined as a neutrocyte count of < 0.50×109/L) showing for at least 48 hours

Exclusion Criteria:

* Age<18 or >80 years old;
* Partial pressure of arterial carbon dioxide (PaCO2) > 50 mmHg or arterial pH < 7.20;
* PaO2/FiO2 >170 or PaO2/FiO2< 85;
* Patients have been treated with NIV or IMV within 30 days.
* NIV is contraindicated or IMV is definitely indicated, including PaO2/FiO2< 85, respiratory arrest, hemodynamic instability, inability to fit the face mask, pneumothorax, vomiting, development of airway bleeding, inability to protect the airway, or copious respiratory secretions;
* Comorbided with other severe diseases, including New York Heart Association functional class ≥ II, valvular heart disease, dilated cardiomyopathy, cardiogenic pulmonary edema, implanted cardiac pacemaker, unstable angina, myocardial infarction, or cardiac surgery within the previous 3 months; systolic arterial pressure <90 mmHg after optimal fluid therapy; history of chronic obstructive pulmonary disease (COPD) or asthma; impaired consciousness (Glasgow Coma Scale score <13); postoperative acute respiratory failure; pregnancy or breastfeeding;
* Lack of consent, do-not-intubate decision, and any other situations where obvious bias are expected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | the 30th day after patient inclusion in the study

SECONDARY OUTCOMES:
In-hospital mortality | through study study completion, an average of 2 years
Length of stay in hospital | through study study completion, an average of 2 years
Length of mechanical ventilation | through study study completion, an average of 2 years
Nosocomial infections | through study study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Li, M.D., Study Chair — PUMC hospital,Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang T, Liu G, He K, Lu X, Liang X, Wang M, Zhu R, Li Z, Chen F, Ke J, Lin Q, Qian C, Li B, Wei J, Lv J, Li L, Gao Y, Wu G, Yu X, Wei W, Deng Y, Wang F, Zhang H, Zheng Y, Zhan H, Liao J, Tian Y, Yao D, Zhang J, Chen X, Yang L, Wu J, Chai Y, Shou S, Yu M, Xiang X, Zhang D, Chen F, Xie X, Li Y, Wang B, Zhang W, Miao Y, Eddleston M, He J, Ma Y, Xu S, Li Y, Zhu H, Yu X. The efficacy of initial ventilation strategy for adult immunocompromised patients with severe acute hypoxemic respiratory failure: study protocol for a multicentre randomized controlled trial (VENIM). BMC Pulm Med. 2017 Sep 20;17(1):127. doi: 10.1186/s12890-017-0467-6. PMID 28931394